CLINICAL TRIAL: NCT07078201
Title: Comparative Analysis of Intraoperative Effect Dexmedetomidine and Fentanyl as an Adjuvant to Heavy Bupivacaine in Spinal Anaesthesia in Lower Limb Orthopedic Surgeries.
Brief Title: Comparative Analysis of Intraoperative Effect Dexmedetomidine and Fentanyl as an Adjuvant to Heavy Bupivacaine in Spinal Anaesthesia in Lower Limb Orthopedic Surgeries to Evaluate the Hemodynamic Stability and Onset and Duration of Motor Block of Using Intrathecal Dexmedetomidine and Fentanyl
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nashwa Ahmed (Other)
Responsible Party: Sponsor-Investigator, Nashwa Ahmed, , Lecturer of Anaesthesia and Surgical Intensive Care, Faculty of Medicine, Port Said University, Egypt, Port Said University hospital
Organization: Port Said University hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB00012098- Serial0307331
Record Dates: First submitted 2025-06-28; First posted 2025-07-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Spinal Anesthesia Duration
MeSH Terms: interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- Group F (Active Comparator)
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — patients received 3 mL volume of 0.5% hyperbaric bupivacaine and 4 µg dexmedetomidine in 0.5 mL of normal saline intrathecal (dexmedetomidine 100 µg/mL diluted in 12.5 ml preservative-free normal saline, 0.5 ml had been withdrawn).
  Arms: Group D
Drug: fentanyl — patients received 3 mL volume of 0.5% hyperbaric bupivacaine with 25 µg fentanyl (0.5 mL) intrathecal.
  Arms: Group F

SUMMARY:
Spinal anesthesia is the most widely employed procedure for lower limb orthopedic operations, as it is very cost-effective and simple to apply. These advantages could be restricted because presently existing local anesthetic drugs had relatively short length of action. (1) Spinal anesthesia with 0.5% heavy bupivacaine (hyperbaric) is a common technique, still there was burden of its short duration of action. To overcome this issue, there was a continuous search for an ideal adjuvant.(2) Adjuvants were mostly added to local anesthetic drugs to increase their effectiveness, speedy onset, increase the period of the block, and reduce the local anesthetics dosage, thus reduction their adverse effects.(3) Such adjuvants had been beneficial in extension of analgesia along with initiation of movement though their related side effects.(4)

DETAILED DESCRIPTION:
Administration of opioids intrathecal such as fentanyl, morphine, and buprenorphine, allowed decreasing dose of the local anesthetic drug, augment analgesic effectiveness, and reduce probable toxicity and cardiovascular adverse consequences of local anesthetics. (5, 2) Nevertheless, adverse effects such as possibly disastrous delayed respiratory depression, urinary retention, nausea, pruritus, vomiting, and constipation had provoked further study to investigate non opioid analgesic drugs with less troublesome drawbacks. (6,2,7,8) Dexmedetomidine is a novel central alpha2-agonist that was approved by the FDA in 1999. It had sedation, anxiolytic, analgesic, and sympatholytic effect that depress cardiovascular reflexes in perioperative interval. (2) Thus, this study had been conducted for assessment of the effectiveness of addition 4 µg Dexmedetomidine to hyperbaric Bupivacaine intrathecally in lower limb orthopaedic surgeries.

Aim This clinical comparative study aimed to evaluate the hemodynamic stability and onset and duration of motor block of using intrathecal dexmedetomidine and fentanyl as an adjuvant to heavy bupivacaine in lower limb orthopaedic surgeries.

Patients and Methods After approval of medical institutional ethical committee, 40 patients of American Society of Anaesthesiologists (ASA) physical status 1or 2, aged between 20-60 years had been incorporated in this prospective randomized controlled study.

Inclusion Criteria

1. The patient aged range from 20 to 60 years 2. ASA 1 and 2 3. Patient prepared for elective lower limb orthopaedic surgeries. 4. Height 150-180 cm. 5. Weight 50-70 kg. 6- Either sex male or female. Exclusion Criteria

1. Patient refusal.
2. Patient had absolute contraindication to spinal anaesthesia.
3. Patients with neurological disorders, pregnancy, local infection at the site of injection.
4. Patients suffering from dysrhythmia or heart block.
5. Patients with ASA 3 or more. An informed written consent had been taken from all the contributors. Patients had been divided into the following groups using randomizer software. Group D: patients received 3 mL volume of 0.5% hyperbaric bupivacaine and 4 µg dexmedetomidine in 0.5 mL of normal saline intrathecal (dexmedetomidine 100 µg/mL diluted in 12.5 ml preservative-free normal saline, 0.5 ml had been withdrawn).

Group F: patients received 3 mL volume of 0.5% hyperbaric bupivacaine with 25 µg fentanyl (0.5 mL) intrathecal.

In preoperative room area: clinical history and examination had been evaluated, and then non-invasive blood pressure and heart rate had been measured and recorded as baseline values.

Anesthetic technique

* Patients would be moved to operation table, 18G IV access was inserted and secured.
* Preloading began15minutes before spinal anaesthesia administration with ringer lactated 20ml /kg.
* Intraoperative monitoring involved NIBP, pulse rate, ECG, SPO2.
* Patients were divided randomly into two groups by using randomizer software.
* Baseline vital signs had been measured. Under strict aseptic technique, after the local infiltration with 2% lignocaine, lumbar puncture was done using 25 G Quincke spinal needle, at L 3 - L 4 space after free flow of csf was verified. Instantly after spinal injection, the patient was placed in a supine position with a cushion supporting shoulders and head. O2 (4-6L/min) had been provided throughout face mask.

The following parameters had been measured: Intraoperatively non-invasive mean blood pressure and heart rate had been documented, every 15 min for first 30minutes then every 30 min till the end of the surgery. onset time of bromage 3 motor block had been recorded (Onset of the motor block; period between the ending of intrathecal drug injection and entire motor paralysis) Duration of motor block had been evaluated by the time taken to return from complete Bromage motor block (bromage 3) to scale 0.

Motor block was evaluated with Modified Bromage scale (6) Bromage 0: The patient could move the hip, knee, and ankle. Bromage 1: The patient could move the hip but had ability to move the knee and ankle.

Bromage 2: The patient could move the hip and knee but had ability to move the ankle.

Bromage 3: The patient could not move the hip, knee, and ankle.

Complications would be noted Intraoperative:

nausea, vomiting, pruritis. Hypotension (> 20% fall of baseline blood pressure or systolic blood pressure of <100mmHg.) had been treated with bolus dose of 6 mg ephedrine IV Bradycardia (pulse rate < 60 bpm), had been treated with 0.3- 0.6 mg atropine IV Incidence of respiratory depression defined as respiratory rate less than 9 /min and SpO2 less than 90% on room air, would be noted, it had been treated with Oxygen (2 L/min), administered via a mask.

ELIGIBILITY:
Inclusion Criteria:

1. The patient aged range from 20 to 60 years
2. ASA 1 and 2
3. Patient prepared for elective lower limb orthopaedic surgeries.
4. Height 150-180 cm.
5. Weight 50-70 kg. 6- Either sex male or female.

Exclusion Criteria:

- 1- Patient refusal. 2- Patient had absolute contraindication to spinal anaesthesia. 3-Patients with neurological disorders, pregnancy, local infection at the site of injection.

4- Patients suffering from dysrhythmia or heart block. 5- Patients with ASA 3 or more.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
to evaluate duration of motor block of using intrathecal dexmedetomidine and fentanyl as an adjuvant to heavy bupivacaine in lower limb orthopedic surgeries. | 7 hour
  Duration of motor block had been evaluated by the time taken to return from complete Bromage motor block (bromage 3) to scale 0.
  Motor block was evaluated with Modified Bromage scale (6) Bromage 0: The patient could move the hip, knee, and ankle. Bromage 1: The patient could move the hip but had ability to move the knee and ankle.
  Bromage 2: The patient could move the hip and knee but had ability to move the ankle.
  Bromage 3: The patient could not move the hip, knee, and ankle.
evaluate onset of motor block of using intrathecal dexmedetomidine and fentanyl as an adjuvant to heavy bupivacaine in lower limb orthopedic surgeries. | 10 minutes
  onset time of bromage 3 motor block had been recorded (Onset of the motor block; period between the ending of intrathecal drug injection and entire motor paralysis)
to evaluate non invasive mean blood pressure using intrathecal dexmedetomidine and fentanyl as an adjuvant to heavy bupivacaine in lower limb orthopedic surgeries. | 90 minutes
  Intraoperatively non-invasive mean blood pressure had been documented, every 15 min for first 30minutes then every 30 min till the end of the surgery.
to evaluate the heart rate using intrathecal dexmedetomidine and fentanyl as an adjuvant to heavy bupivacaine in lower limb orthopedic surgeries. | 90 minutes
  Intraoperatively heart rate had been documented, every 15 min for first 30minutes then every 30 min till the end of the surgery.

SECONDARY OUTCOMES:
Complications would be noted Intraoperative | 90 minutes
  nausea, vomiting, pruritis. Hypotension (> 20% fall of baseline blood pressure or systolic blood pressure of <100mmHg.) had been treated with bolus dose of 6 mg ephedrine IV Bradycardia (pulse rate < 60 bpm), had been treated with 0.3- 0.6 mg atropine IV Incidence of respiratory depression defined as respiratory rate less than 9 /min and SpO2 less than 90% on room air, would be noted, it had been treated with Oxygen (2 L/min), administered via a mask.

CONTACTS AND LOCATIONS:
Locations (1):
- Port said university, Port Said, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gupta R, Verma R, Bogra J, Kohli M, Raman R, Kushwaha JK. A Comparative study of intrathecal dexmedetomidine and fentanyl as adjuvants to Bupivacaine. J Anaesthesiol Clin Pharmacol. 2011 Jul;27(3):339-43. doi: 10.4103/0970-9185.83678. PMID 21897504
- [Result] Rajasekaran S, Murugaih S, Anandan A, Ramalingam A. A comparative study of intrathecal clonidine VS dexmedetomidine in caesarean patients. Indian Journal of Clinical Anaesthesia 2018;5(1):68-74.
- [Result] Sharma E, Gupta B, Verma RK, Devra V. Block characteristics of different doses of intrathecal dexmedetomidine when combined with low dose heavy bupivacaine for gynecological surgeries: a double blind, randomised comparative study. Sch. J. App. Med. Sci., 2017; 5(6D):2286-2294.
- [Result] Ahmed SA, Lotfy HA, Mostafa TAH. The effect of adding dexmedetomidine or dexamethasone to bupivacaine-fentanyl mixture in spinal anesthesia for cesarean section. J Anaesthesiol Clin Pharmacol. 2024 Jan-Mar;40(1):82-89. doi: 10.4103/joacp.joacp_396_22. Epub 2024 Mar 14. PMID 38666154
- [Result] Gupta A, Gupta KL, Yadav M. To evaluate the effect of addition of dexmedetomidine to hyperbaric bupivacaine intrathecally in infraumblical surgeries. International Journal of Contemporary Medical Research 2016;3(7):2136-2138.
- [Result] Kumar S, Choudhury B, Varikasuvu SR, Singh H, Kumar S, Lahon J, Saikia D. A Systematic Review and Meta-analysis of Efficacy and Safety of Dexmedetomidine Combined With Intrathecal Bupivacaine Compared to Placebo. Cureus. 2022 Dec 12;14(12):e32425. doi: 10.7759/cureus.32425. eCollection 2022 Dec. PMID 36644042
- [Result] Reddy NG, Sekar RG, Ahmed CJ, Himabindu M, Mallika CH, Tejaswini PK. Intrathecal nalbuphine versus dexmedetomidine as an adjuvant in spinal anaesthesia for lower limb and lower abdominal surgeries. Journal of Cardiovascular Disease Research 2023;14(2): 825-883.
- [Result] Zhang Y, Shan Z, Kuang L, Xu Y, Xiu H, Wen J, Xu K. The effect of different doses of intrathecal dexmedetomidine on spinal anesthesia: a meta-analysis. Int J Clin Exp Med 2016;9(10):18860-18867.

DOCUMENTS (1):
  • Study Protocol (2025-06-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT07078201/Prot_000.pdf